CLINICAL TRIAL: NCT03987035
Title: Physician-Initiated Trial Investigating the BeGraft Peripheral Stent Graft System as Bridging Stent in FEVAR for Complex Aortic Aneurysms
Brief Title: BGP Stent as Bridging Stent in FEVAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marc Bosiers, MD (Other)
Responsible Party: Sponsor-Investigator, Marc Bosiers, MD, Director, FCRE (Foundation for Cardiovascular Research and Education)
Organization: FCRE (Foundation for Cardiovascular Research and Education) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCRE-200504
Record Dates: First submitted 2019-06-12; First posted 2019-06-14 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Thoracoabdominal Aortic Aneurysm, Without Mention of Rupture; Abdominal Aortic Aneurysm, Without Mention of Rupture
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal; Aortic Aneurysm, Abdominal

STUDY DESIGN:
Intervention Model Description: Application of BeGraft Peripheral Stent Graft System as bridging stent in Fenestrated Endovascular Repair (FEVAR) for complex aortic aneurysms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BGP Stent Graft System (Experimental): BGP Stent Graft System as bridging stent in Fenestrated Endovascular Repair (FEVAR) for complex aortic aneurysms
  Interventions: Device: BeGraft Peripheral (BGP) Stent Graft System as bridging stent

INTERVENTIONS:
Device: BeGraft Peripheral (BGP) Stent Graft System as bridging stent — BGP Stent Graft System as bridging stent
  Other Names: implant of stent graft BGP

SUMMARY:
The objective of this clinical investigation is to evaluate, in a controlled setting, the safety and performance of the BeGraft Peripheral (BGP) balloon expandable covered stent Graft System (Bentley InnoMed, Hechingen, Germany) implanted as bridging stent in FEVAR (fenestrated endovascular aortic repair) for complex aortic aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for elective repair of AAA/TAAA extent IV with FEVAR in accordance with the applicable guidelines for vascular interventions (Aneurysm size 5.5cm or aneurysm growth of >5 mm within 6 months or 1 cm within 1 year).
* Patient is willing to comply with specified follow-up evaluations at the specified times
* Patient is >55 years old
* Patient understands the nature of the procedure and provides written informed consent, prior to enrollment in the study
* Patient has a projected life-expectancy of at least 12-months
* Indication of elective repair of AAA or TAAA with FEVAR in accordance with the applicable guidelines for vascular interventions
* Patient needs to have a landing zone in their target vessel of at least 10mm
* No early important division branch from the target vessel with risk of coverage
* Absence of dissection
* Target vessels (renal arteries, superior mesenteric artery and celiac trunk) should have a diameter between 5 and 10 mm
* Patient eligible for fenestrated endovascular repair as per IFU of the fenestrated endograft
* Angulation of the aorta at the level of the target vessels <45 degrees
* The fenestrated endograft has to be constructed so the fenestrations lie in front of the orifice of the target vessel, and the gap between the fenestration and the orifice of the target vessel should not exceed 10mm.

Exclusion Criteria:

* Previously implanted endograft
* Patients refusing treatment
* Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated
* Patients with uncorrected bleeding disorders or heparin induced thrombozytopenia
* Female patient with child bearing potential not taking adequate contraceptives or currently breastfeeding
* Any planned surgical intervention/procedure within 30 days of the study procedure
* Any patient considered to be hemodynamically unstable at onset of procedure
* Patient is currently participating in another investigational drug or device study that has not completed the entire follow up period.
* Patients with diffuse distal disease resulting in poor stent outflow
* Fresh thrombus formation
* Stenosed (>50%) or occluded target vessel
* Angulation between renal artery and aortic wall <30 degrees
* Patients with known hypersensitivity to the stent material (L605) and/or PTFE
* Hybrid Approach
* Patients with a connective tissue disorder
* Patients with mycotic or inflammatory aneurysm
* Myocardial infarction or stroke within 3 months prior to the procedure
* Patients with an unstable angina pectoris or heart insufficiency NYHA 3 or 4
* Patients with ASA classification 5 or higher
* Contraindications against contrast enhanced angiography (a.e. massive hyperthyroidism)
* Patients with increased risk of intraoperative rupture
* Patients with access vessel which are too tortuous, narrow or any kind of reason that would lead to failure of introducing and advancing an introducer sheath

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Efficacy endpoint (1) - Technical success | 1 day post-op
  Successful introduction and deployment of the BeGraft Peripheral (BGP) balloon expandable covered stent Graft System (Bentley Innomed, Hechingen, Germany) implanted as bridging stent in FEVAR
Efficacy endpoint (2) ) Bridging stent patency at 12 months | 12 months post-op
  defined as absence of restenosis (≥50% stenosis) or sole target vessel occlusion based on CT Angio at 12 months
Safety endpoint at 12 months | 12 months post-op
  Absence of procedure related complications and bridging stent related endoleaks at 12 months

SECONDARY OUTCOMES:
Bridging stent patency post-procedure | 1 day post-op, 6-, 12, and 24- months post-op
  Bridging stent patency post-op and at 6-, 12- and 24-months, defined as absence of restenosis (≥50% stenosis) or sole target vessel occlusion based on Duplex ultrasound or CT Angio
Freedom from bridging stent related endoleaks post-procedure | 1 day post-op, 6-, 12, and 24- months post-op
  Freedom from bridging stent related endoleaks post-op and at 6-, 12- and 24- months, based on imaging (duplex ultrasound, CT angiography)
Freedom from bridging stent related secondary intervention post-procedure | 1 day post-op, 6-, 12, and 24- months post-op
  Freedom from bridging stent related secondary intervention post-op, 6-, 12- and 24- months
Freedom from type I & III endoleaks post-procedure | 1 day post-op, 6-, 12, and 24- months post-op
  Freedom from type I & III endoleaks post procedure and at 6, 12 and 24-months, based on imaging (duplex ultrasound, CT angiography)
30-day mortality | 30 days post-op
Freedom from stent graft migration post-procedure | 1 day post-op, 6-, 12, and 24- months post-op
  defined as freedom from stent graft migration (more than 10 mm)
Freedom from AAA diameter increase | 6-, 12, and 24- months post-op
  defined as more than 5mm increase in maximum diameter measured at 6- , 12- and 24- months as compared to postop-implantation, based on imaging (duplex ultrasound or CT Angiography)
Freedom from aneurysm related secondary endovascular procedures post-procedure | 1 day post-op, 6-, 12, and 24- months post-op
  Freedom from aneurysm related secondary endovascular procedures
Freedom from conversion to open surgical repair post-procedure | 1 day post-op, 6-, 12, and 24- months post-op
  Freedom from conversion to open surgical repair post-op
Freedom from aneurysm related mortality post-procedure | 1 day post-op, 6-, 12, and 24- months post-op
  Freedom from aneurysm related mortality post-procedure
Freedom from aneurysm rupture within 12- and 24-months post-implantation | 12, and 24- months post-op
  Freedom from aneurysm rupture within 12- and 24-months post-implantation
Freedom from any major adverse events post-procedure | 1 day post-op, 6-, 12, and 24- months post-op
  Freedom from any major adverse events post-procedure
Health Related Quality of Life scores | 12- and 24-months post-op
  Health Related Quality of Life scores at 12- and 24-months post implantation

CONTACTS AND LOCATIONS:
Overall Officials: Eric Verhoeven, Prof. Dr., Principal Investigator — Foundation for Cardiovascular Research and Education
Locations (9):
- Germany (9):
  - Alexander Gombert, Aachen
  - University Heart Center Freiburg- Bad Krozingen, Freiburg im Breisgau
  - University Hospital Gießen, Giessen
  - University Hospital Hamburg-Eppendorf, Hamburg
  - University Hospital LMU Munich, München
  - Martin Austermann, Münster
  - Klinikum Nürnberg Süd, Nuremberg
  - University Hospital Regensburg, Regensburg
  - Hospital Stuttgart, Stuttgart

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Bentley announces FEVAR indication for BeGraft and launch of new BeFlared fenestrated bridging stent - Vascular News — https://vascularnews.com/bentley-announces-fevar-indication-for-begraft-and-launch-of-new-beflared-fenestrated-bridging-stent/